CLINICAL TRIAL: NCT06146660
Title: CAMZYOS® (Mavacamten) Post-Marketing Surveillance in Korean Patients With Symptomatic Obstructive Hypertrophic Cardiomyopathy (oHCM)
Brief Title: A Study to Assess the Safety of Mavacamten in Korean Patients With Symptomatic Obstructive Hypertrophic Cardiomyopathy
Status: Recruiting | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CV027-1089
Record Dates: First submitted 2023-11-15; First posted 2023-11-27 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Obstructive Hypertrophic Cardiomyopathy
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic | interventions — MYK-461

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants receiving mavacamten for oHCM
  Interventions: Drug: Mavacamten

INTERVENTIONS:
Drug: Mavacamten — According to approved product label

SUMMARY:
The purpose of this observational post-marketing surveillance study is to assess the real-world safety of mavacamten for the treatment of symptomatic obstructive hypertrophic cardiomyopathy (oHCM) in adult participants in Korea. Participants who will receive at least 1 dose of mavacamten will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants 19 years of age or older
* Participants who receive mavacamten according to the approved product label
* Participants who sign the informed consent form

Exclusion Criteria:

* Participants who are prescribed mavacamten for therapeutic indications not approved in Korea
* Participants for whom mavacamten is contraindicated as clarified in Korean prescribing information approved by the Ministry of Food and Drug Safety

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants diagnosed with symptomatic oHCM who will receive mavacamten according to the approved product label
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2024-07-24 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events | Up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (2):
- South Korea (2):
  - Local Institution - 0001, Seoul
  - Novotech Laboratory Korea Co., Ltd., Seoul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html